CLINICAL TRIAL: NCT03400735
Title: Comparison of Cefdinir and Cefdinir/Clavulanic Acid Combination in Treatment of Acute Exacerbation of Chronic Bronchitis (AECB) and Community-acquired Pneumonia (CAP) in Adults
Brief Title: Comparison of Cefdinir and Cefdinir/Clavulanic Acid Combination in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-08.16
Record Dates: First submitted 2016-10-03; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Acute Exacerbation of Chronic Bronchitis; Community-Acquired Pneumoniae
MeSH Terms: interventions — Cefdinir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefdinir/clavulanic acide 300/125 mg Film Coated Tablets (Experimental)
  Interventions: Drug: Cefdinir 300Mg Capsule
- Cefdinir 300 mg Capsules (Active Comparator)
  Interventions: Combination Product: Cefdinir/clavulanic acide 300/125 mg film-coated tablets

INTERVENTIONS:
Combination Product: Cefdinir/clavulanic acide 300/125 mg film-coated tablets — Cefdinir is already an approved drug. In this study, developed cefdinir/clavulanic acide combination will be compared against to cefdinir alone.
  Other Names: Fullcef Plus
  Arms: Cefdinir 300 mg Capsules
Drug: Cefdinir 300Mg Capsule — Cefdinir is used as comparator
  Arms: Cefdinir/clavulanic acide 300/125 mg Film Coated Tablets

SUMMARY:
It is planned to compare the efficacy and safety of cefdinir and cefdinir/clavulanic acide treatments in acute exacerbation of chronic bronchitis (AECB) and community-acquired pneumoniae (CAP) patients.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of chronic bronchitis
* The diagnosis of community-acquired pneumoniae
* FEV1 value = 30-80%
* The diagnosis of mild-severe acute exacerbation of chronic bronchitis (AECB)
* Oxygen saturation < 90%

Exclusion Criteria:

* Pregnancy or breastfeeding
* Allergy against to penicillin or cephalosporins
* Renal impairment
* Active hepatic disease
* Antibiotic use except study drugs
* Immunosuppressive therapy before 6 months of study initiation
* Use of probenecid like drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
The comparison of clinical success rates according to laboratory parameters | 7-10 days

SECONDARY OUTCOMES:
The comparison of remission or relief of inflammation according to laboratory parameters | 7-10 days
The comparison of patient satisfaction according to satisfaction questionnaire | 7-10 days
The comparison of adverse events | 7-10 days

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Erzincan University Mengücek Gazi Training and Research Hospital, Erzincan
  - Yedikule Chest Diseases Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided